CLINICAL TRIAL: NCT03660267
Title: The Effects of Coffee Ingestion on Recovery of Bowel Function in Patients Undergoing Benign Gynecologic Operation : A Randomized Controlled Trial
Brief Title: >The Purpose of This Study Was to Determine Whether Consuming a 100-mL Cup of Coffee is Effective in Preventing or Reducing Postoperative Ileus After Laparotomy of Benign Gynecological Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: coffeeaof
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2018-07

CONDITIONS: Effects of Coffee Ingestion on Recovery of Bowel Function
Keywords: Benign Gynecologic Operation; Coffee Ingestion; Recovery of Bowel Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- coffee group (Experimental): caffeine coffee
  Interventions: Other: caffeine coffee
- decaffeinete coffee group (Experimental): decaffeinete coffee group
  Interventions: Other: decaffiene coffee
- water group (Experimental)
  Interventions: Other: still water

INTERVENTIONS:
Other: caffeine coffee — drank 3 cups of caffeinated coffee daily (100 mL at 05:00 AM, 10:00 PM, and 15:00 PM), beginning on the morning after surgery Patients were free to drink any amount of water but no more coffee, black tea, or other form of caffeine, such as soda.
  Coffee was prepared with a conventional coffee machine
  Arms: coffee group
Other: decaffiene coffee — drank 3 cups of decaffeinated coffee daily (100 mL at 05:00 AM, 10:00 PM, and 15:00 PM), beginning on the morning after surgery Patients were free to drink any amount of water but no more coffee, black tea, or other form of caffeine, such as soda.
  Coffee was prepared with a conventional coffee machine
  Arms: decaffeinete coffee group
Other: still water — drank 3 cups of still water daily (100 mL at 05:00 AM, 10:00 PM, and 15:00 PM), beginning on the morning after surgery Patients were free to drink any amount of water but no more coffee, black tea, or other form of caffeine, such as soda.
  Coffee was prepared with a conventional coffee machine
  Arms: water group

SUMMARY:
Comparison of the effectiveness coffee (with or without caffeine) ingestion and water for reducing the duration of Postoperative ileus after Laparotomy of Benign Gynecological Patients

DETAILED DESCRIPTION:
laparotomy benign gynecological surgery is the most common gynecologic operation worldwide because is major operation for surgery and can affect to bowel movement after operation and turn to postoperative ileus , clinically severe postoperative ileus affects up to 14% of patients after laparotomy for gynecologic surgery that leaded to more complication, slowly recovery , prolong length of hospitalized stay and consequently increase unnecessary cost of treatment.

Preclinical studies has considered to use preventative therapeutic options for prevent ileus including coffee

The investigators used the coffee reduces postoperative ileus However, no good quality of evidence base supports the effectiveness coffee (with or without caffeine) ingestion and water for reducing the duration of Postoperative ileus after Laparotomy of Benign Gynecological Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients were asked to participate if they were scheduled to undergo laparotomy for a benign gynecologic condition
* Ever drink coffee before
* can speak or communication Thai language

Exclusion Criteria:

1 hypersensitivity or allergy to caffeine/ coffee 2.ever intraabdominal sugery before 3. had an active intra-abdominal malignancy, bowel perforation, pre-existing bowel disease, or a history of abdominal or pelvic irradiation.

4.pregnancy woman 5.thyroid disease 6 Inflammatory bowel disease 7.liver disease 8.cardiac arrhythmia 9.history of difficult to defecation ( feces only 2 times per week) 10.after operation need to stay in ICU more than 24 hr 11.need to put Ng tube after operation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
time to flatus | ึ7 day
  measure time to first flatus after finished operation

SECONDARY OUTCOMES:
time to toleration of a solid diet | 7 day
  The time to tolerance of a solid diet was measured from the end of surgery (defined as when the patients woke up from anesthesia) until the patient tolerated the intake of solid food (any food that required chewing) without vomiting or experiencing significant nausea within 4 hours after the meal and without reversion to enteral fluids only
time to defecation | 7 day
  measure time to first defecation after finished operation

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Phaya Thai, Bangkok, Thailand